CLINICAL TRIAL: NCT00579982
Title: An Open-Label Trial Measuring Satisfaction and Convenience of Two Formulations of Lamotrigine in Subjects With a Mood Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBI108884
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Mood Disorders
Keywords: Mood disorder
MeSH Terms: conditions — Mood Disorders | interventions — Lamotrigine

ARMS (1):
- Arm 1 (Experimental): Lamictal orally disintegrating tablet (ODT)
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Experimental formulation

SUMMARY:
To determine the convenience and satisfaction of new orally disintegrating tablet formulation (ODT) of lamictal in subjects with a mood disorder. This was a multicenter, open-label study in participants with a mood disorder, who reported difficulty or discomfort in swallowing the currently marketed IR compressed tablet formulation of lamotrigine and who had a person (such as a spouse, partner, companion, aid, nurse, caregiver, etc) willing to complete a Companion/Caregiver Question. Subjects were switched from the currently marketed lamotrigine IR formulation to a matching dose of lamotrigine IR orally disintegrating tablet (ODT) for 3 weeks to determine convenience and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a documented diagnosis of a mood disorder as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV (296.00-296.90).
* Subject must have a person (such as a spouse, partner, companion, aid, nurse, caregiver, etc) willing to complete a Companion/Caregiver Preference Question either in person or via the telephone. This individual must read, write, and comprehend English at a level sufficient to complete study-related assessments.
* Subject must have been taking a stable dose of currently marketed compressed tablet formulation of lamotrigine IR for at least 4 weeks prior to Baseline (Day 1) of the study and must be adherent to the prescribed dosing regimen. The current dose must not exceed 600 mg/day.
* Subject's current lamotrigine IR dose, frequency and number of tablets per administration must remain consistent between the IR and ODT regimens. However, the subject's current lamotrigine IR dose may be such that the subject would receive no more than one additional ODT per administration in order to equal their IR dose.
* Subject must currently report a difficulty or discomfort swallowing lamotrigine IR compressed tablets, the nature of which is or will be documented. NOTE: A diagnosis of dysphagia is not required.
* Subject must have the ability to comprehend the consent form and provide informed consent.
* Subject must read, write, and comprehend English at a level sufficient to complete study-related assessments.
* Subject is a male or female at least 18 years of age.
* If female, the subject is eligible to enter and participate in this study if she is not lactating and is of:

  1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is pre-menarchal or post-menopausal [defined as one year without menses]); is surgically sterile [via hysterectomy and/or removal of the ovaries] or,
  2. child-bearing potential, has a negative pregnancy test at both Screening and/or Baseline (prior to Investigational Product administration), and agrees to one of the following requirements:
* has a male sexual partner who is surgically sterilized (vasectomy with documentation of azoospermia) prior to Screening or,
* sexual partner(s) is/are exclusively female or,
* double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository). The subject must be using this method for at least 1 week following the discontinuation of Investigational Product or,
* any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year. Acceptable IUDs, for the purposes of this study, include TCu-380A (Paragard), TCU-380 Slimline (Gyne T Slimline), MULTILOAD-250 (MLCu-250) and 375, Levonorgesterol LNG-20 Intrauterine System (Mirena/Levonova), and Flexigard 330/CuFix PP330 (Gynefix).The subject must have had the device inserted at least 2 weeks prior to Screening, throughout the study, and 2 weeks following the discontinuation of Investigational Product.

Exclusion Criteria:

* Subject has:
* a current (or within six months prior to Screening) diagnosis of anorexia nervosa or bulimia.
* a diagnosis of a mood disorder due to a general medical condition, or substance abuse per DSM-IV (293.83).
* a diagnosis of schizophrenia or other psychotic disorders.
* Subject who meets current criteria of an acute mood disorder and has a CGI-S of ≥4 at Screening.
* Subject who crushes lamotrigine IR compressed tablet prior to taking or receiving medication orally.
* Subject who, in the investigator's judgment, poses a homicidal or serious suicidal risk; has made a suicide attempt within the six months preceding Screening; or has ever been homicidal.
* Subject who has a score of 1 or greater on Suicidality item (Item 9) of the BDI-II at Screening and/or Baseline.
* Subject has ever experienced a rash related to prior lamotrigine treatment, or for whom treatment was discontinued for clinically significant safety reasons.
* Subject has a history of severe hepato-biliary disease within the past 3 years.
* Subject has any medical condition that, in the investigator's judgment, is considered to be clinically significant and could potentially affect subject safety or study outcome.
* Subject has a positive urine test at Screening for illicit drug use and/or a history of alcohol or substance abuse or dependence within the past 12 months.
* Subject is currently participating in another clinical study in which the subject is or will be exposed to an investigational or non-investigational drug or device, or has done so within the preceding month for studies unrelated to the current illness, or six months for studies related to the current illness.
* Female subject is pregnant, lactating, or does not agree to use contraceptive method(s) specified in the protocol to avoid pregnancy during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- United States (17):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Orange City, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Fairview Heights, Illinois
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Olean, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Sajatovic M, Thompson TR, Nanry K, Edwards S, Manjunath R. Prospective, open-label trial measuring satisfaction and convenience of two formulations of lamotrigine in subjects with mood disorders. Patient Prefer Adherence. 2013 May 7;7:411-7. doi: 10.2147/PPA.S40271. Print 2013. PMID 23687443
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: LBI108884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LBI108884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LBI108884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LBI108884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LBI108884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LBI108884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LBI108884 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine: Orally Disintegrating Tablet (ODT). ODT dosing was to match the dose and regimen of the immediate release (IR) dose the subject was taking at baseline. The mean (standard deviation [SD]) ODT dose was 261.3 (118.9) mg/day.
Period: Overall Study
Arm/Group | Lamotrigine
Started | 97
Completed | 89
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.07)
Gender [Count of Participants; unit: Participants]
  Female | 83
  Male | 14
Race/Ethnicity, Customized [Number; unit: participants]
  White | 94
  Black | 2
  Mixed race | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Convenience Subscale Score (CSS) Derived From the Treatment Satisfaction Questionnaire for Medication (TSQM v 1.4) Using Items 9 (Ease of Use), 10 (Ease of Planning to Use), and 11 (Convenience) at Week 3.
Description: The CSS is the sum of items 9 (values: 1=Extremely difficult - 7=Extremely easy), 10 (same set of values as for 9), and 11 (1=Extremely inconvenient - 7=Extremely convenient). The sum has 3 subtracted from it, is divided by 18, and then multiplied by 100; the range is 0-100. Change from baseline=end of study CSS minus baseline score.
Time Frame: Baseline, End of Study (Week 3) or Early Withdrawal
Population: Intent to Treat (ITT). Ninety-eight participants were enrolled in the study, but one withdrew prior to receiving lamotrigine ODT treatment. All efficacy and safety analyses are based on the Intent to Treat population, which includes the 97 patients who received at least one dose of ODT treatment.
Measure: Mean (Standard Deviation); unit: Points on a subscale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Points on a subscale | 23.3 (22.5)
Statistical Analysis 1: Comparison: Lamotrigine; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Paired t-test

2. Secondary Outcome: Mean Change From Baseline in the Global Satisfaction Subscale Score, From the TSQM Using Items 12 (Confidence in Medicine), 13 (Certainty That Good Things About Medication Outweigh Bad Things), and 14 (Satisfaction With Medication) at Week 3
Description: The Global Satisfaction Subscale Score is the sum of item 12 (values: 1=Not at all confident - 5=Extremely confident), item 13 (values: 1=Not at all certain - 5=Extremely certain), and item 14 (Extremely dissatisfied - 7=Extremely satisfied). The sum has 3 subtracted from it, is divided by 14, and then multiplied by 100; thus, the range is 0-100.
Time Frame: Baseline, End of Study (Week 3) or Early Withdrawal
Population: ITT
Measure: Mean (Standard Deviation); unit: Points on a subscale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Points on a subscale | -0.3 (29.34)

3. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression of Illness-Severity at Week 3
Description: Clinician assessment evaluating how mentally ill the patient is at time of evaluation. The questionnaire is based on a 7-point scale (from1 = Normal to 7 = Among the most extremely ill patients).
Time Frame: Baseline, End of Study (Week 3) or at Early Withdrawal
Population: ITT
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 96
Points on a scale | 0.0 (0.81)

4. Secondary Outcome: Mean Change From Baseline in the Beck Depression Inventory (BDI-II) Score at Week 3
Description: Participant-reported questionnaire consisting of 21 items on a 4 point scale (0 to 3, with 3 indicating most severely ill), with the score being the sum of the items. The change from baseline is the end of study score minus the baseline score; larger values indicate more depression with the ODT formulation relative to the IR formulation.
Time Frame: Baseline, End of Study (Week 3 weeks) or at Early Withdrawal
Population: ITT
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Points on a scale | -1.7 (9.52)

5. Secondary Outcome: Number of Participants Answering the Question "Did the Tablets Dissolve Instantly (Yes or no)?" at Week 3
Description: The Organoleptic Questionnaire (9 items) was used to assess the participants' satisfaction with the physical characteristics of the ODT formulation e.g. rate of dissolution, flavor. Question number 1 on organoleptic questionnaire: Did the tablets dissolve instantly (yes or no)?
Time Frame: End of Study (Week 3) or Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  Yes | 60
  No | 37

6. Secondary Outcome: Number of Participants Answering the Question "How Satisfied or Dissatisfied Were You With the Time it Took the Tablet to Dissolve" at Week 3
Description: Question number 2 on organoleptic questionnaire: How satisfied or dissatisfied were you with the time it took the tablet to dissolve? [from a rating of 1 (Extremely dissatisfied) to 5 (Extremely satisfied)]
Time Frame: Baseline, End of Study (Week 3) or Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  Extremely dissatisfied | 3
  Very dissatisfied | 10
  Satisfied | 37
  Very satisfied | 18
  Extremely satisfied | 29

7. Secondary Outcome: Number of Participants Answering the Question "How Did the Dissolved Tablet Feel in Your Mouth?" at Week 3
Description: Question number 3 on organoleptic questionnaire: How did the dissolved tablet feel in your mouth? [from a rating of 1 (Extremely gritty) to 5 (Extremely smooth)]
Time Frame: End of Study (Week 3) or Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  Extremely gritty | 0
  Very gritty | 19
  Smooth | 45
  Very smooth | 19
  Extremely smooth | 14

8. Secondary Outcome: Number of Participants Answering the Question "How Satisfied Were You With the Flavor of the Tablet?" at Week 3
Description: Question number 4 on organoleptic questionnaire: How satisfied were you with the flavor of the tablet? [from a rating of 1 (Extremely dissatisfied) to 5 (Extremely satisfied)]
Time Frame: End of Study (Week 3) or Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  Extremely dissatisfied | 5
  Very dissatisfied | 10
  Satisfied | 26
  Very satisfied | 23
  Extremely satisfied | 33

9. Secondary Outcome: Number of Participants Answering the Question "How Would You Rate the Strength of the Flavor of the Tablet"? at Week 3
Description: Organoleptic Questionnaire, question 5: How would you rate the strength of the flavor of the tablet? [from 1 a rating of (Extremely bothersome) to 5 (Extremely pleasant)]
Time Frame: End of Study (Week 3) or Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  Extremely bothersome | 2
  Very bothersome | 14
  Pleasant | 36
  Very pleasant | 22
  Extremely pleasant | 23

10. Secondary Outcome: Number of Participants Answering the Question "How Would You Rate the Aftertaste of the Tablet"? at Week 3.
Description: Organoleptic Questionnaire, question 6: How would you rate the aftertaste of the tablet (the taste remaining in your mouth after swallowing the tablet)? [from a rating of 1 (Extremely bothersome) to 6 (Did NOT experience an aftertaste)]
Time Frame: End of Study (Week 3) or Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  Extremely bothersome | 4
  Very bothersome | 20
  Pleasant | 25
  Very pleasant | 7
  Extremely pleasant | 12
  I did NOT experience an aftertaste | 29

11. Secondary Outcome: Number of Participants Answering the Question "How Satisfied Were You With the Aftertaste of the Tablet"? at Week 3
Description: Organoleptic Questionnaire, question 7: How satisfied were you with the aftertaste of the tablet (the taste remaining in your mouth after swallowing the tablet)? [from a rating of 1 (Extremely dissatisfied) to 6 (I did NOT experience an aftertaste)]
Time Frame: Baseline, End of Study (Week 3) or Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  Extremely dissatisfied | 3
  Very dissatisfied | 16
  Satisfied | 28
  Very satisfied | 11
  Extremely satisfied | 11
  I did NOT experience an aftertaste | 28

12. Secondary Outcome: Number of Participants Answering the Question "Compared to Standard Tablets That Need to be Swallowed With Liquid, How Convenient or Inconvenient Did You Find This Orally Disintegrating Tablet"? at Week 3
Description: Organoleptic Questionnaire, question 8: Compared to standard tablets that need to be swallowed with liquid, how convenient or inconvenient did you find this orally disintegrating tablet? (from a rating of 1 [Extremely inconvenient] to 5 [Extremely convenient])
Time Frame: End of Study (Week 3) or at Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  Extremely inconvenient | 8
  Very inconvenient | 9
  Convenient | 16
  Very convenient | 17
  Extremely convenient | 47

13. Secondary Outcome: Number of Participants Answering the Question "Compared to Standard Tablets That Need to be Swallowed With Liquid, How Easy or Difficult is it to Use This Orally Disintegrating Tablet?" at Week 3
Description: Organoleptic Questionnaire, question 9: Compared to standard tablets that need to be swallowed with liquid, how easy or difficult is it to use this orally disintegrating tablet? [from a rating of 1 (Extremely difficult) to 5 (Extremely easy)]
Time Frame: End of Study (Week 3) or at Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  Extremely difficult | 2
  Very difficult | 3
  Easy | 17
  Very easy | 20
  Extremely easy | 55

14. Secondary Outcome: Number of Participants Indicating a Preference for ODT or the Standard IR Tablet at Week 3
Description: Participant indicated whether preference was for ODT or the standard IR tablet
Time Frame: End of Study (Week 3) or at Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  Prefer ODT | 72
  Prefer standard IR tablet | 25

15. Secondary Outcome: Number of Companions/Caregivers Indicating Whether ODT or Standard IR Tablet is More Convenient at Week 3
Description: Companion/Caregiver indicates whether ODT is more convenient or standard IR tablet is more convenient
Time Frame: End of Study (Week 3) or at Early Withdrawal
Population: ITT
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 97
Number of participants
  ODT more convenient | 79
  Standard IR tablet more convenient | 18

16. Secondary Outcome: Number of Participants Indicating at Week 3 (by Answering Yes/no) That They Would be More Likely to Take the ODT Formulation
Description: Tablet Routine Questionnaire (Adherence): Adherence to the treatment was evaluated by asking if the participant would be more likely to take the ODT formulation (yes/no)
Time Frame: End of Study (Week 3) or at Early Withdrawal
Population: ITT: Only 94 of the 97 subjects in the ITT Population responded to the Tablet Routine Questionnaire.
Measure: Number; unit: Number of participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 94
Number of participants
  Yes | 84
  No | 10

ADVERSE EVENTS:
Arm/Group | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 1/97
Other Adverse Events (participants affected / at risk) | 28/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine (N=97)
Myocardial infarction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine (N=97)
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Hypomania (Psychiatric disorders) | 3
Depressed mood (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastrooeophageal reflux disease (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Chest pain (General disorders) | 1
Influenza-like illness (General disorders) | 1
Irritability (General disorders) | 1
Pain (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Vision blurred (Eye disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.